CLINICAL TRIAL: NCT01625364
Title: Comparison of Asthma Programs for Schools
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Eileen K. Kintner, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01NR010544-05 (NIH)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Asthma; Reactive Airway Disease
Keywords: Health Education; Health Counseling; Patient Education
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Health Education | interventions — Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Airways for Schools (Experimental): OAS is a school-based non-academic asthma health education program for elementary students with asthma and their parents.
  Interventions: Behavioral: Open Airways for Schools
- SHARP program (Experimental): The Staying Health-Asthma Responsible & Prepared (SHARP) program is an academic and counseling asthma health education program for older school-age students with asthma and members of their social networks including their family caregiver.
  Interventions: Behavioral: SHARP program

INTERVENTIONS:
Behavioral: SHARP program — Staying Healthy-Asthma Responsible and Prepared is an academic and counseling asthma health education program for older school-age students with asthma and members of their social networks including their family caregivers.
  Other Names: Staying Healthy-Asthma Responsible and Prepared
  Arms: SHARP program
Behavioral: Open Airways for Schools — OAS is a non-academic asthma health education program for elementary students with asthma and their parents.
  Other Names: OAS
  Arms: Open Airways for Schools

SUMMARY:
The purpose was to evaluate effectiveness and impact of an academic and counseling asthma health education program (SHARP) for fourth- and fifth-grade students diagnosed with asthma. Students attending schools randomized to the low-dose control condition received Open Airways for Schools (OAS). The first aim was to evaluate the effectiveness of SHARP, compared to the low-dose group, for students on cognitive, psychosocial, and behavioral aspects of asthma management at 1, 12, and 24 months post-intervention. We hypothesized that compared to students enrolled in elementary schools who received the low-dose program, students in elementary schools that received SHARP would increase asthma knowledge (cognition) and logical reasoning abilities for managing acute episodes (cognition), acceptance of asthma as a chronic condition (psychosocial), and use of effective asthma health behaviors (behavior). The second aim was to evaluate the long-term impact of SHARP, compared to the low-dose group, for students on condition characteristics, use of healthcare services, and quality of life at 12 and 24 months post intervention. We hypothesized that compared to students enrolled in elementary schools who received the low-dose program; students in elementary schools who received SHARP would decrease asthma severity, use of healthcare services, and school absenteeism due to asthma, and increase participation in life activities (quality of life).

DETAILED DESCRIPTION:
Over 7 million US children younger than age 18 years are currently diagnosed with asthma, and approximately 4 million children experience exacerbation of asthma symptoms annually. The NIH National Guidelines for the Diagnosis and Management of Asthma specify that part of a successful management program includes educating students with asthma and their caregivers about the condition. The guidelines recommend expanding education of students and families to schools and community settings. An academic and counseling program was developed for older school-age students with asthma and their family caregivers titled Staying Healthy-Asthma Responsible & Prepared™ (SHARP). A two-group prospective randomized single-blinded design was used. The sample consisted of two cohorts of students diagnosed aged 9-12 years with asthma and their caregivers from varying socioeconomic, racial, and ethnic backgrounds. Cohort dyads were drawn from 23 elementary schools that were located in a diverse, moderately sized, medically underserved, inner-city community. The schools were matched based on projected enrollment numbers, standardized reading and math scores, free/reduced lunch eligibility, and racial/ethnic proportions prior to randomization. Recently retired certified elementary schoolteachers, identified by the district, were trained to serve as interveners to deliver both programs in the schools during instructional time.

ELIGIBILITY:
Inclusion Criteria:

* Student eligibility inclusion criteria included (a) a diagnosis of asthma, (b) availability to participate in scheduled classes or make-up sessions, and (c) verbal and written assent to participate in the study. Caregiver eligibility inclusion criteria included (a) being a caregiver of a student with asthma, (b) ability to understand English, and (c) expressed availability to attend and participate in the community program.

Exclusion Criteria:

* Exclusion criteria included student's expressed unwillingness to participate or lack of consent from parent/legal guardian. Severity of symptoms was not a criterion for eligibility. Exclusion criteria included expressed unwillingness to participate or lack of consent.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reasoning about Asthma Management | 24 months or 2 years post-intervention
  Evidence of statistically significant increase in older school-age student reasoning about managing symptom exacerbation during an acute asthma episode.

SECONDARY OUTCOMES:
Participation in Life Activities | 24 months or 2 years post-intervention
  Evidence of statistically significant improvement in quality of life as evidenced by increase in participation in life activities score.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen K Kintner, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States